CLINICAL TRIAL: NCT03110393
Title: Prospective Randomized Comparison Between a Fiber Optic Intubation Via the Ambu® AuraGain ™ or the i-Gel® Laryngeal Mask Until a Complete Airway Protection in Obese Patients
Brief Title: Ambu®AuraGain™ Versus I-gel® in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Berthold Moser, Principal Investigator, Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_10
Record Dates: First submitted 2017-03-20; First posted 2017-04-12 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Obese
Keywords: Obese; Laryngeal Mask Airway; Anaesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu® AuraGain™ (Experimental): Intervention with Ambu® AuraGain™Laryngeal Mask
  Interventions: Device: Ambu AuraGain
- Intersurgical i-gel® (Active Comparator): Intervention with Intersurgical i-gel® Laryngeal Mask
  Interventions: Device: Intersurgical i-gel

INTERVENTIONS:
Device: Ambu AuraGain — Insert and intubation of an Ambu® AuraGain™ laryngeal mask
  Arms: Ambu® AuraGain™
Device: Intersurgical i-gel — Insert and intubation of an Intersurgical i-gel®
  Arms: Intersurgical i-gel®

SUMMARY:
The aim of this study is the randomized comparison of two laryngeal mask (Intersurgical i-gel® and Ambu®AuraGain™) in obese patients

DETAILED DESCRIPTION:
Since the incidence of a difficult intubation lies between 4.5% -7.5%, the search for alternative airway devices has been forced in the past.

As an option, the laryngeal mask is suitable, which has been used as a universal airway with a high degree of safety in routine anesthesia.

There are numbers of different laryngeal masks available which have the characteristic to insert an endotracheal tube through the ventilation lumen.

The indications for these laryngeal masks can be extended due to continuous improvements in the laryngeal masks, these laryngeal masks can also be used in obese patients. Obese patients generally have a 4-fold increased risk of a difficult airway, and a BMI over 35 is a predictor of a difficult tracheal intubation.

There are no studies comparing the Intersurgical i-gel® Laryngeal Mask and the Ambu®AuraGain ™ Laryngeal Mask in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Shoulder-/Elbow-/Hip-/Knee- or Foot - Surgery
* Signed informed consent
* BMI > 35kg/m2

Exclusion Criteria:

* Non-sober patients (last meal <6 h)
* Symptomatic reflux disease
* Hiatus hernia
* Significant cardiovascular risk factors
* Severe COPD
* Gastric band or gastric bypass
* Disease which allows an accurate examination of the physicians (e.g. neuromuscular, mental, metabolic disease)
* Drug or drug abuse in the recent past
* Legal immaturity (incompetence)
* Acute disease, which calls into question the narcotic potential
* Patients with whom the use of a laryngeal mask is contraindicated or otherwise not possible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Time of successful intubation | intraoperative
  Measurement of a fiberoptic intubation with the laryngeal mask. Start: Insertion of the fiberoptic into the larynxmask until the intubation has been done and after the fiberoptic has been removed.

SECONDARY OUTCOMES:
Number of Insertions (of the laryngeal mask) | intraoperative
  Number of insertion attempts will be registered
Time of insertion | intraoperative
  The time of Insertion of the laryngeal mask will be recorded.
Number of insertion attempts | intraoperative
  Number of insertions with the stomach tube will be registered
Gastric volume | intraoperative
  Measurement of the gastric volume
Positioning of the gastric probe | intraoperative
  Determination of the position of the gastric probe after successful insertion by stethoscope.
Successful Ventilation | intraoperative
  Detection of a successful Ventilation. There are two options: a tidal volume > 6mL/kg lean body mass or endtidal pCO2 < 6.7kPa
Oropharyngeal leak pressure of the Ambu®AuraGain ™ | intraoperative
  The oropharyngeal leak pressure of the AuraGain™ is measured with a measured cuff volume of 60cmH2O
Oropharyngeal leak pressure of the Intersurgical i-gel® | intraoperative
  The oropharyngeal leak pressure of the Intersurgical i-gel® is measured.
Measurement of blood pressure | intraoperative
  Measurement of blood pressure during 5min (1 measurement / minute).
Measurement of oxygen saturation | intraoperative
  Measurement oxygen saturation during 5min (1 measurement / minute).
Measurement of heart rate | intraoperative
  Measurement of heart rate during 5min (1 measurement / minute).
Maximum ventilation pressure | intraoperative
  The maximum ventilation pressure is measured, which must be applied in order to adequately ventilate the patients. This is measured over 5 minutes
Measurement CO2 (kPa): | intraoperative
  The exhaled CO2 is determined continuously.
Number of intubation attempts | intraoperative
  The number of intubation attempts until successful intubation is recorded.
Reasons for the unsuccessful intubation | intraoperative
  The reasons are listed in tabular form.
Number of esophageal intubations | intraoperative
  The number of esophageal intubations is measured.
Resistance (for an EET): | intraoperative
  The resistance is measured with a score of 1- 4. 1: simple passage, no resistance, 2: little resistance for the passage, 3: significant resistance for the passage, 4: passage not possible
Location of the mask (Brimacombe) | intraoperative
  The position of the mask is determined by pushing the fiber optic to a maximum of 1cm over the LMA and then using the Brimacombe score.
Swallowing (no / little / medium / strong) | 5hour postoperative
  The swallowing difficulties are questioned preoperatively and postoperatively (5 (± 1) h after anesthesia end).
Throat pain (no / little / medium / strong) | 5hour postoperative
  The throat pain is questioned preoperatively and postoperatively (5 (± 1) h after anesthesia end).
Hoarseness (no / little / medium / strong) | 5hour postoperative
  The swallowing difficulties, the throat pain and the hoarseness are questioned preoperatively and postoperatively (5 (± 1) h after anesthesia end).
Blood on laryngeal mask after intubation | intraoperative
  Determination of the visible blood on the laryngeal mask after removal (no, little, much).

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Berthold, MD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moser B, Keller C, Audige L, Dave MH, Bruppacher HR. Fiberoptic intubation of severely obese patients through supraglottic airway: A prospective, randomized trial of the Ambu(R) AuraGain laryngeal mask vs the i-gel airway. Acta Anaesthesiol Scand. 2019 Feb;63(2):187-194. doi: 10.1111/aas.13242. Epub 2018 Aug 8. PMID 30088266